CLINICAL TRIAL: NCT03320655
Title: Effectiveness of Combined Aerobic and Strength Training in Acute and Chronic Adaptations in Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Maria Helena Santa-Clara Pombo Rodrigues, Assistant Teacher, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 28/2017
Record Dates: First submitted 2017-10-16; First posted 2017-10-25 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Chronic Heart Failure; Fragility
Keywords: Chronic Heart Failure; Fragility

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Aerobic Training (Active Comparator): The subjects will perform in ST part, always only 1 set in the 6 machines early mentioned. During the first and second week they will do 12 repetitions at 40% - 50% of 1 RM. In the third and fourth week progress to 10 repetitions at 60%-70% of 1 RM, and in the second and third month, 8 repetitions at 70%-80% of 1 RM. In the AT part the HIIT protocol is based on a ratio 2 min : 1 min. Consisted of 10 interval training periods (2 min of high intensity at 85% - 90% of heart rate reserve (HRreser) and 9 pauses (1 min in passive pause) between interval training periods. During the first week of training will start with a continuous training, in the second week will start with 5 intervals of HIIT, and in the second and third months they are doing the 10 stages of HIIT.
  Interventions: Other: Combined Strength Training
- Combined Strength Training (Experimental): During the first and second week subjects will perform 1 sets with 12 repetitions at 40% - 50% of 1 RM in the 6 machines mentioned before. In the third and fourth week strength exercises progress to 2 sets of 10 repetitions, at 60%-70% of 1 RM, and in the second and third month consists of 3 sets at 8 repetitions, at 70%-80% of 1 RM. In the AT part the HIIT protocol is based on a ratio 2 min : 1 min. Consisted of of 5 interval training periods (2 min of high intensity: 85% - 90% of HRreser) and 4 pauses (1 min in passive pause) between interval training periods. During the first week of training will start with a continuous training, in the second week will start with 3 intervals of HIIT, and after the third/fourth week they are doing the 5 stages of HIIT.
  Interventions: Other: Combined Aerobic Training

INTERVENTIONS:
Other: Combined Aerobic Training — The subjects will perform in ST part, always only 1 set in the 6 machines early mentioned. During the first and second week they will do 12 repetitions at 40% - 50% of 1 RM. In the third and fourth week progress to 10 repetitions at 60%-70% of 1 RM, and in the second and third month, 8 repetitions at 70%-80% of 1 RM. In the AT part the HIIT protocol is based on a ratio 2 min : 1 min. Consisted of 10 interval training periods (2 min of high intensity at 85% - 90% of heart rate reserve (HRreser) and 9 pauses (1 min in passive pause) between interval training periods. During the first week of training will start with a continuous training, in the second week will start with 5 intervals of HIIT, and in the second and third months they are doing the 10 stages of HIIT.
  Arms: Combined Strength Training
Other: Combined Strength Training — During the first and second week subjects will perform 1 sets with 12 repetitions at 40% - 50% of 1 RM in the 6 machines mentioned before. In the third and fourth week strength exercises progress to 2 sets of 10 repetitions, at 60%-70% of 1 RM, and in the second and third month consists of 3 sets at 8 repetitions, at 70%-80% of 1 RM. . In the AT part the HIIT protocol is based on a ratio 2 min : 1 min. Consisted of of 5 interval training periods (2 min of high intensity: 85% - 90% of HRreser) and 4 pauses (1 min in passive pause) between interval training periods. During the first week of training will start with a continuous training, in the second week will start with 3 intervals of HIIT, and after the third/fourth week they are doing the 5 stages of HIIT.
  Arms: Combined Aerobic Training

SUMMARY:
Patients with chronic heart failure (CHF) underwent to a hospital-based cardiac rehabilitation (CR) program in the Lisbon district Hospitals will be recruited. The participants will be randomized into one of the following exercise groups: A) combined exercise training with more aerobic training and less strength training (CAT); B) combined exercise training with more strength training and less aerobic training (CST). The investigators will test two proportions in combined training, CAT and CST. There hasn't been any data on the so called combined regimes, which include both aerobic exercise with HIIT and ST and the investigators will evaluate the effects of acute and chronic response.

The research project will contribute to a better understanding in several aspects that are unexplained by scientific research.

DETAILED DESCRIPTION:
Literature Review:CHF is the major public health problem in the world[1], highly prevalent in older individuals and a major cause of disability, hospitalizations, morbidity and mortality[2]. Generally, CHF patients have reduced exercise capacity, with main symptoms of effort intolerance, early fatigue and breathlessness[3], also exhibiting increased peripheral and central chemosensitivity, and impaired sympathovagal balance with sympathetic activation(SA) predominance[4].

Understanding the oxidative metabolism and intracellular energy transfer in both skeletal and cardiac muscle, mechanisms of endothelial dysfunction, and the role of SA and inflammatory cytokines provide possible mechanistic explanations of the pathophysiologic factors involved in the development of exercise intolerance[5,6]. It has been shown in CHF patients that increased arterial stiffness is associated with cardiovascular morbidity and mortality[7]. There are evidences that increased arterial stiffness predicts exercise intolerance in CHF patients[8].

Increased carotid IMT is associated with subclinical left ventricular(LV) myocardial dysfunction, suggesting a possible role of carotid IMT in HF risk determination [9]. CHF is associated too with endothelial dysfunction including impaired endothelium-mediated, flow-dependent dilation(FMD). Since endothelial function is thought to play an important role in coordinating tissue perfusion and modulating arterial compliance, interventions to improve endothelial dysfunction are imperative.

Systemic vasoconstriction and impaired peripheral perfusion are hallmarks in advanced CHF. While a number of factors, including increased sympathetic tone and an activated renin-angiotensin system, have been proposed to be involved in the reduced arterial vasodilatory capacity in HF, the pivotal role of the endothelium in coordinating tissue perfusion has now been recognized.

Several clinical studies have documented endothelial dysfunction of large conduit and small resistance vessels in patients with CHF. Endothelial dysfunction may affect the cardiovascular system in two ways: first, endothelial dysfunction of resistance vessels may impair peripheral perfusion, and, second, endothelial dysfunction of large conduit vessels may limit the increase in blood flow provided by the supplying large vessels and may increase impedance of the failing LV and consequently impair LV ejection fraction(LVEF). An important functional consequence of endothelial dysfunction is the inability to release nitric oxide(NO) in response to physiological stimuli such as increases in flow, reflecting impaired FMD[10]. Conversely, chronically increased blood flow enhances the release of NO in experimental models, by upregulation of NO synthase, the enzyme that uses L-arginine to generate NO. The intermittent increases of blood flow by physical training may increase the capability of the endothelium to release NO and therefore may restore endothelial function in patients with CHF who are usually subjected to a limited degree of physical activity[5]. The dysfunctional endothelium contributes to increased vascular stiffness and impaired arterial distensibility, augmenting myocardial damage[10].

The direct relationship between exercise and vascular health is certain, but the complex set of metabolic pathways, haemodynamic effects of exercise on cardiovascular cells/tissues, and the regulation of genetic expression activated by exercise is still largely undefined[11]. The effects of aerobic and resistance exercise on clinical blood pressure might be different, because they have different mechanical characteristics. Aerobic training(AT) is characterized by the execution of cyclic exercises, carried out with large muscle groups contracting at mild to moderate intensities for a long period of time. On the other hand, strength training(ST) is characterized by the execution of exercises in which muscles from a specific body segment are contracted against a force that opposes the movement[12].

Aerobic capacity is directly related to arterial function, including endothelial function, arterial stiffness and wave reflection. In addition, coupling of arterial and cardiac function is a major determinant of aerobic capacity. Thus, poor resting arterial function likely limits aerobic capacity, but it is also possible that changes in arterial function during acute exercise may play a role. Arterial function is not only associated with aerobic capacity, but is also an independent predictor of mortality[5].

Controlled clinical trials have shown that in HF patients ExT programs improve peripheral and cardiac adaptations and also the aerobic capacity, delay the onset of anaerobic metabolism, and improve the autonomic balance[1,13]. Apart from adaptation in maximal cardiac output, heart contractility, and stroke volume, aerobic ExT is also able to promote amelioration in the peripheral microvascular background by reducing resistance to flow, increasing the compliance of the arteries and endothelial function [13]. Abnormalities in endothelium and FMD are a key phenomenon in the blunted vasodilatory response in CHF patients. ExT enables the improvement of both basal endothelial NO formation and agonist-mediated FMD of the skeletal muscle(SM) vasculature in CHF patients. The correction of endothelial dysfunction is associated with a significant improvement in exercise capacity evidenced by a 26% increase in peak oxygen uptake(VO2peak)[14].

Previous studies in HF have been showing that 16.4% of 171 patients had cachexia, and the mortality at 18 months of follow up was as high as 50% in the subset of patients with cachexia compared with 17% in those without cachexia. Cardiac cachexia is defined as an advanced stage of HF associated with involuntary loss of at least 5% of non-oedematous body weight. And muscle wasting, also known as sarcopenia, is the loss of muscle mass(MM) and strength, whereas cachexia describes loss of weight. Distinction of the two clinical conditions might also be challenging, because cachexia and muscle wasting can co-exist in the same patient. Indeed, cachexia might lead to muscle wasting and vice versa, although muscle wasting can occur earlier in the course of the disease[15].

SM strength, in upper and lower limbs, are parameters that independently predict survival[16,17,18]. This alternative treatment should focus on increasing MM, strength and power in the limbs to improve functionality and performance[19]. SM dysfunction includes reduced cardiac contractile performance that contributes to changes in SM physiology, muscle atrophy, weakness and reduced oxidative capacity [20]. Muscle function is also enhanced in response to ST in CHF patients, including myofilament function and whole muscle[21] as well as SM oxidative capacity[21].

It's crucial that the ExT in such patients should be train the peripheral muscles effectively without producing great cardiovascular stress. An alternative treatment approach should focus on the application of specific resistance exercise program to improve body composition[22], increase the cross-sectional area, muscle fiber[23], all of which counteract muscle wasting and may be cornerstone in the prevention of sarcopenia and cardiac cachexia in CHF patients[24].

ExT is a major component of rehabilitation/secondary prevention interventions, inducing significant beneficial changes in mechanisms of pathophysiology, exercise tolerance, functional capacity and QoL, while a positive impact on hospitalization and mortality reduction. There has been growing interest in the characteristics and modalities of exercise training able to induce optimal benefits. High intensity and interval mode have been shown to induce greater benefits than moderate intensity and continuous mode regimes. Considering the current body of evidence of high-intensity interval training(HIIT) in CHF, HIIT demonstrated to be more efficient, resulting in long-term adherence, which be an important practical aspect to consider during the ExT and consequently optimized improvements in central and peripheral adaptations[25]. More studies are needed to proof their safety and benefits on this type of patients.

Additionally, there has been sound rationale for the inclusion of ST to the HIIT, which has been also shown able to yield benefits in terms of exercise capacity and QoL. It is well known that combined AT and ST is the preferred exercise intervention to reverse or attenuate the loss of MM and improve exercise and functional capacity, muscle strength in this individuals[19]. But there are underlying mechanisms from the ST in the CHF patient's peripheral capacity that remains unidentified. And isn't known what is the benefits of combine different proportions of AT and ST.

For that reason, the investigators will test two proportions in combined training, CAT and CST. There hasn't been any data on the so called combined regimes, which include both aerobic exercise with HIIT and ST and the investigators will evaluate the effects of acute and chronic response.

Purpose:The research project will contribute to a better understanding in several aspects that are unexplained by scientific research. The purpose of this research project are:

1. To determine the effectiveness of an ExT programme with different proportions of CAT and CST in promoting cumulative effects in acute and chronic adaptations in CHF patients;
2. To identify the mechanisms of the potential improvement in effectiveness promoted by ST; This research project is going to employ state of the art methods focusing peripheral adaptations analysis in both groups namely in echocardiography variables, cardiopulmonary exercise testing, arterial stiffness, functional physical fitness, QoL and body composition in 2 distinguished moments: M1)baseline and M2)3 month.

Plan and Methods:This project will assess the acute and chronic effects in central and peripheral adaptations of a combined training to patients with CHF would address a number of important breaches in scientific knowledge with potential clinical benefits.

Study Design: A longitudinal randomized control trial (RCT) research design using two distinct ExT prescriptions (CAT and CST) will be applied in CHF patients. All the same assessments will be done in two moments: M0 - baseline and M1 - 3 months after starting the ExT. The patients will be randomized into either one of the two ExT group.

Recruitment and screening will last 9 months(October 2017 to June 2018) and the patient assessment will last until August 2018. It is expected to finish the project with peer-review redaction submitted and/or accepted in December 2018.

The following assessments on the 4 moments will be performed at the host Hospital, FMH-UL: Echocardiogram(Echo); cardiopulmonary exercise test(CPET); arterial stiffness - Complior Analyse; Intima-media thickness - ultrasound; body composition - dual-energy radiographic absorptiometry; functional physical fitness - Fullerton Functional Fitness Test; isometric strength - portable hand dynamometer JAMAR plus digital; maximal strength - 1RM and QoL questionnaire.

All assessment moments will be done in 4 days:

Day 1-The CPET, Echo will be performed at the host Hospital; Day 2 and 3-during one day and time of the ExT session at the host hospital, the patient will perform the functional physical fitness tests; maximal strength; isometric strength and QoL questionnaire. In another day the investigators will perform the arterial stiffness and the IMT before the session in rest and after the ExT; Day 4-In FMH, and dual-energy radiographic absorptiometry(DXA) exam. Individual reports will be sent by email or delivered on paper. During the 1-year project the multidisciplinary team will have bimonthly meetings to update the study information and discuss the patient's progress.

ELIGIBILITY:
Inclusion Criteria:

* CHF patients; receiving optimal medical therapy for CHF (including an angiotensin-converting enzyme inhibitor or an angiotensin receptor blocker and a beta-blocker unless a contraindication is evident) with a stable condition for more than 1 month (no hospitalization for heart failure (HF), no change in medication, and no change in New York Heart Association (NYHA) functional class.

Exclusion Criteria:

* If they are younger than 18 years or are unable to sign informed consent; unstable angina pectoris; and orthopedic or neurological limitations to exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Echocardiogram at 3 months | At baseline and 3 months after Cardiac Rehabilitation
  A resting transthoracic echocardiogram will be performed with MyLab Alpha, ESAOTE, Italy. The exam will be performed by the echocardiography laboratory cardiologists, who will be blinded to experimental protocol and group randomization, with the usual measurements of systolic and diastolic function, particularly the calculation of LVEF by Simpson's formula, telediastolic and telessystolic volumes and diameters, doppler analysis of the transmitral flow, tissue doppler and quantification of mitral valve regurgitation.
Change from Baseline Cardiopulmonary Exercise Test at 3 months | At baseline and 3 months after Cardiac Rehabilitation
  This test will be performed with the subjects in a non-fasting condition and under the regular medication.
  A symptom-limited ramp incremental CPET, will be performed on a cycle ergometer with breath-by-breath gas exchange measurements. Each patient will be encouraged to exercise to exhaustion. Patients will continue seated on the cycle ergometer as soon as they stop, while recovery measurements are taken. Blood pressure will be continuous recorded Peak oxygen capacity will be considered the highest attained VO2 during the final 30 sec of exercise and ventilator AT will be estimate by the V-slope method. The recovery period will continue until 6 min after peak effort. All patients should achieve a respiratory exchange ratio of >1.1.
  We will study, the HR max and recovery at 1st and 3rd min, the VO2 peak, respiratory exrespiratory exchange ratios, respiratory quotient, ventilatory anaerobic threshold, the ventilatory equivalent for O2 and CO2 .
Change from Baseline Arterial Stiffness at 3 months | At baseline and 3 months after Cardiac Rehabilitation
  Arterial stiffness will be measured by pulse wave velocity(PWV) obtained by applanation tonometry will be measured during a 15 and 30min rest.A single operator locates the arteries on the right side of the body and mark the point for capturing the corresponding pressure curves with 2 specific pressure sensitive transducers. The distance between the carotid and femoral, radial and distal posterial tibial arteries will be measured directly and entered into the Complior Analyse software. Right brachial blood pressure will be measured and entered in software, and then signal acquisition is launched. When the operator observes 10 carotid pulse wave forms of at least90% quality showed on the software, pressure curves will be recorded. Values obtained from the carotid to femoral artery, carotid to radial artery and carotid to distal posterial tibial artery are taken as indices of central/aortic, upper and lower limb arterial stiffness, respectively.
Change from Baseline Intima-Media Thickness at 3 months | At baseline and 3 months after Cardiac Rehabilitation
  Carotid intima media thickness(cIMT) will be defined as the distance between the leading edge of the lumen-intima interface to the leading edge of the media-adventitia interface of the far wall of the right carotid artery using an ultrasound scanner. cIMT is automatically measured, and distension curves are acquired within a segment of the carotid artery about 1cm before the flow divider, where the operator places the region of interest.
  To evaluate the acute effects of ExT, at the pre-exercise measurement at 5,15and 30min rest, blood pressure(BP) was measured twice on the right upper arm in a dorsal decubitus position. The final measured value was used for the analysis. Immediately after measuring BP. Post-exercise measurement was carried out with the same methods.
  From this test, the investigators will study the diameter and distensibility of the artery,cIMT, PWV, brachial blood pressure, and the alpha and beta index.
Change from rest Arterial Stiffness and post effort | Assessment before session in 15 minutes rest and after session at 5, 15 and 30 minutes pos effort
  Arterial stiffness will be measured by pulse wave velocity(PWV) obtained by applanation tonometry will be measured during a 15 and 30min rest.A single operator locates the arteries on the right side of the body and mark the point for capturing the corresponding pressure curves with 2 specific pressure sensitive transducers. The distance between the carotid and femoral, radial and distal posterial tibial arteries will be measured directly and entered into the Complior Analyse software. Right brachial blood pressure will be measured and entered in software, and then signal acquisition is launched. When the operator observes 10 carotid pulse wave forms of at least90% quality showed on the software, pressure curves will be recorded. Values obtained from the carotid to femoral artery, carotid to radial artery and carotid to distal posterial tibial artery are taken as indices of central/aortic, upper and lower limb arterial stiffness, respectively.
Change from rest Intima-Media Thickness and post effort | Assessment before session in 15 minutes rest and after session at 5, 15 and 30 minutes pos effort
  Carotid intima media thickness(cIMT) will be defined as the distance between the leading edge of the lumen-intima interface to the leading edge of the media-adventitia interface of the far wall of the right carotid artery using an ultrasound scanner. cIMT is automatically measured, and distension curves are acquired within a segment of the carotid artery about 1cm before the flow divider, where the operator places the region of interest.
  To evaluate the acute effects of ExT, at the pre-exercise measurement at 5,15and 30min rest, blood pressure(BP) was measured twice on the right upper arm in a dorsal decubitus position. The final measured value was used for the analysis. Immediately after measuring BP. Post-exercise measurement was carried out with the same methods.
  From this test, the investigators will study the diameter and distensibility of the artery,cIMT, PWV, brachial blood pressure, and the alpha and beta index.

SECONDARY OUTCOMES:
Change from Baseline Body Composition- Dual Energy Radiographic at 3 months ABSORPTIOMETRY | At baseline and 3 months after Cardiac Rehabilitation
  All the patients will be tested in the morning with a 12h fasted no caffeine and alcohol, refrained from the moderate to vigorous exercise at least 24h. Total and regional body mass is estimated using dual energy radiographic absorptiometry(DXA). This technique uses RX with a low radiation dose(1-3μSv/test), much lower than usual exposure to our natural involvement(5-8μSv/day) or RX to the chest (50-150μSv / test). Total body skeletal muscle mass(TBSMM) will be calculated as TBSMM=(1.13 ALST)-(0.02 age)+(0.61 sex)+0.97, where ALST means appendicular lean soft tissue. Skeletal muscle mass will be normalized by height and termed skeletal muscle index to verify the level of physical disability risk. All anthropometric procedures will be led by the same certified technician.
  We will study the bone mineral content, lean soft- tissue and fat mass, total and regional body mass.
Change from Baseline Objective Measured Physical Activity at 3 months | At baseline and 3 months after Cardiac Rehabilitation
  Each participant will use the ActiGraphGT3X+ and given oral and written instructions on how to wear the accelerometers for the following 7days. The ActiGraph GT3X+ is able to assess acceleration in the vertical, antero-posterior and medio-lateral axes. The ActiGraph GT3X+ will be attached to an elastic waist belt and placed in line with the axillary line of the right iliac crest. Participants will be asked to wear the accelerometer from the moment they wake up until they go to bed at night, and requested to remove it only during water-based activities such as showering and swimming and when they go to bed. ActiGraphGT3X+ will be initialized using a sample rate of 30Hz and then downloaded using the low filter extension option in Actilife5 Software.The cut off points previously used in an older sample of adults to calculate daily times in each activity intensity band. All physical activity variables will be converted to time (in min) per valid day.
Change from Baseline Funtional Physical Fitness Tests at 3 months | At baseline and 3 months after Cardiac Rehabilitation
  The functional physical fitness tests are a simple, reproducible tool to assess submaximal functional capacity. The 6min walking test will be performed indoors, along a long flat, 20meter corridor. Patients will be instructed to walk at their own pace, with rest stops as needed. The result will be the distance in meters covered in the 6min. The 30sec chair stand,assesses the lower body strength.Patients will be instructed to sit and stand as faster as they can in 30sec with arms folded across chest.The 8-foot(2.4meters) up and go test evaluates the agility, will be evaluated the time in sec that the participant needed to get up, walk the distance of2.44meters and return to the initial position. The chair sit-and-reach aim to assess the lower body flexibility and to assess the upper body flexibility, it will be used the back scratch test.
Change from Baseline Isometric Strength at 3 months | At baseline and 3 months after Cardiac Rehabilitation
  Handgrip strength will be assessed by a portable hand dynamometer JAMAR plus digital. Subjects will be assessed on both hands alternately. Handgrip assessment will be conducted with the patients in a seated comfortable position, with the shoulder adducted and close to, but not supported by, the trunk. The elbow of the assessed limb should be flexed to 90degrees and the forearm should be in a neutral position (halfway between supine and pronation position). A variation of 0-30 degrees in the wrist extension will be allowed. Each subject will be assessed in three attempts for both hands alternately. In each attempt the subject will exert the maximal grip strength on the hand dynamometer with the assessed limb during 5 seconds. After each attempt, there will be a resting period of 60sec that will be used both for recovery and for changing the handgrip dynamometer to the opposite hand. All patients will be instructed not to perform a Valsalva manoeuvre during the tests.
Change from Baseline Maximal Strength at 3 months | At baseline and 3 months after Cardiac Rehabilitation
  Maximal strength will be assessed by 1RM test for each of 6weight exercises on variable resistance machines, leg press, leg extension, leg curl, low row, chest press and lat pull down. Correct exercise and breathing techniques (avoidance of the Valsalva manoeuvre) will be practiced. To warm-up before using a machine, each patient will be asked to perform eight repetitions using a relatively light resistance, followed by a 30sec rest. A second set of 4repetitions using a moderate resistance will be then used, followed by a 1min rest. After that each patient will be asked to perform single repetitions until the 1RM was reached. The rests between attempts will be 1-2min. The resistance will be increased by approximately 5kg, or by 2.5kg when the subject was near his maximum. Strength will be recorded as the maximal number of kilograms lifted in 1 full range of motion.
Change from Baseline Quality of Life Questionnaire at 3 months | At baseline and 3 months after Cardiac Rehabilitation
  The Short Form-36 Health Survey(SF-36) is a self-assessment health status questionnaire composed of 36 questions about socio-demographic, health and personal behavior. It was designed for use in clinical practice and research, health policy evaluations and general population surveys. The 36 questions capture the subject's perception of their general health by sorting them into multi-item scales that assess 8 concepts. The 8 subscales are as follows: physical functioning; role/physical; bodily pain; general health; vitality/energy; social functioning; role/emotional; mental health/emotional wellbeing. The SF-36 also provides 2important summery measures of health-related QoL:physical component summary and mental component summary scales.The strength of both scales lies in their ability to distinguish a physical from a mental outcome. The items and dimensions in SF-36 were constructed using the likert method of summated ratings. A Portuguese validated version of SF-36 is available.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Helena Santa-Clara Pombo Rodrigues, PhD, Principal Investigator — University of Lisbon
Locations (1):
- Faculty of Human Kinetics, Lisbon, Portugal

REFERENCES:
- [Background] Belardinelli R, Georgiou D, Cianci G, Purcaro A. 10-year exercise training in chronic heart failure: a randomized controlled trial. J Am Coll Cardiol. 2012 Oct 16;60(16):1521-8. doi: 10.1016/j.jacc.2012.06.036. Epub 2012 Sep 19. PMID 22999730
- [Background] Loncar G, Fulster S, von Haehling S, Popovic V. Metabolism and the heart: an overview of muscle, fat, and bone metabolism in heart failure. Int J Cardiol. 2013 Jan 10;162(2):77-85. doi: 10.1016/j.ijcard.2011.09.079. Epub 2011 Oct 7. PMID 21982619
- [Background] Tabet JY, Meurin P, Driss AB, Weber H, Renaud N, Grosdemouge A, Beauvais F, Cohen-Solal A. Benefits of exercise training in chronic heart failure. Arch Cardiovasc Dis. 2009 Oct;102(10):721-30. doi: 10.1016/j.acvd.2009.05.011. Epub 2009 Sep 15. PMID 19913773
- [Background] Caldwell JH, Link JM, Levy WC, Poole JE, Stratton JR. Evidence for pre- to postsynaptic mismatch of the cardiac sympathetic nervous system in ischemic congestive heart failure. J Nucl Med. 2008 Feb;49(2):234-41. doi: 10.2967/jnumed.107.044339. Epub 2008 Jan 16. PMID 18199620
- [Background] Downing J, Balady GJ. The role of exercise training in heart failure. J Am Coll Cardiol. 2011 Aug 2;58(6):561-9. doi: 10.1016/j.jacc.2011.04.020. PMID 21798416
- [Background] Belardinelli R. Arrhythmias during acute and chronic exercise in chronic heart failure. Int J Cardiol. 2003 Aug;90(2-3):213-8. doi: 10.1016/s0167-5273(02)00576-4. PMID 12957754
- [Background] Kitzman DW, Herrington DM, Brubaker PH, Moore JB, Eggebeen J, Haykowsky MJ. Carotid arterial stiffness and its relationship to exercise intolerance in older patients with heart failure and preserved ejection fraction. Hypertension. 2013 Jan;61(1):112-9. doi: 10.1161/HYPERTENSIONAHA.111.00163. Epub 2012 Nov 12. PMID 23150511
- [Background] Ooi H, Chung W, Biolo A. Arterial stiffness and vascular load in heart failure. Congest Heart Fail. 2008 Jan-Feb;14(1):31-6. doi: 10.1111/j.1751-7133.2008.07210.x. PMID 18256567
- [Background] Effoe VS, Rodriguez CJ, Wagenknecht LE, Evans GW, Chang PP, Mirabelli MC, Bertoni AG. Carotid intima-media thickness is associated with incident heart failure among middle-aged whites and blacks: the Atherosclerosis Risk in Communities study. J Am Heart Assoc. 2014 May 9;3(3):e000797. doi: 10.1161/JAHA.114.000797. PMID 24815496
- [Background] Marti CN, Gheorghiade M, Kalogeropoulos AP, Georgiopoulou VV, Quyyumi AA, Butler J. Endothelial dysfunction, arterial stiffness, and heart failure. J Am Coll Cardiol. 2012 Oct 16;60(16):1455-69. doi: 10.1016/j.jacc.2011.11.082. Epub 2012 Sep 19. PMID 22999723
- [Background] Whyte JJ, Laughlin MH. The effects of acute and chronic exercise on the vasculature. Acta Physiol (Oxf). 2010 Aug;199(4):441-50. doi: 10.1111/j.1748-1716.2010.02127.x. Epub 2010 Mar 26. PMID 20353494
- [Background] Cardoso CG Jr, Gomides RS, Queiroz AC, Pinto LG, da Silveira Lobo F, Tinucci T, Mion D Jr, de Moraes Forjaz CL. Acute and chronic effects of aerobic and resistance exercise on ambulatory blood pressure. Clinics (Sao Paulo). 2010 Mar;65(3):317-25. doi: 10.1590/S1807-59322010000300013. PMID 20360924
- [Background] Acanfora D, Scicchitano P, Casucci G, Lanzillo B, Capuano N, Furgi G, Acanfora C, Longobardi M, Incalzi RA, Piscosquito G, Ciccone MM. Exercise training effects on elderly and middle-age patients with chronic heart failure after acute decompensation: A randomized, controlled trial. Int J Cardiol. 2016 Dec 15;225:313-323. doi: 10.1016/j.ijcard.2016.10.026. Epub 2016 Oct 11. PMID 27750131
- [Background] Hambrecht R, Fiehn E, Weigl C, Gielen S, Hamann C, Kaiser R, Yu J, Adams V, Niebauer J, Schuler G. Regular physical exercise corrects endothelial dysfunction and improves exercise capacity in patients with chronic heart failure. Circulation. 1998 Dec 15;98(24):2709-15. doi: 10.1161/01.cir.98.24.2709. PMID 9851957
- [Background] von Haehling S, Ebner N, Dos Santos MR, Springer J, Anker SD. Muscle wasting and cachexia in heart failure: mechanisms and therapies. Nat Rev Cardiol. 2017 Jun;14(6):323-341. doi: 10.1038/nrcardio.2017.51. Epub 2017 Apr 24. PMID 28436486
- [Background] Casas-Vara A, Santolaria F, Fernandez-Bereciartua A, Gonzalez-Reimers E, Garcia-Ochoa A, Martinez-Riera A. The obesity paradox in elderly patients with heart failure: analysis of nutritional status. Nutrition. 2012 Jun;28(6):616-22. doi: 10.1016/j.nut.2011.10.006. Epub 2012 Jan 20. PMID 22261572
- [Background] Hulsmann M, Quittan M, Berger R, Crevenna R, Springer C, Nuhr M, Mortl D, Moser P, Pacher R. Muscle strength as a predictor of long-term survival in severe congestive heart failure. Eur J Heart Fail. 2004 Jan;6(1):101-7. doi: 10.1016/j.ejheart.2003.07.008. PMID 15012925
- [Background] Anker SD, Ponikowski P, Varney S, Chua TP, Clark AL, Webb-Peploe KM, Harrington D, Kox WJ, Poole-Wilson PA, Coats AJ. Wasting as independent risk factor for mortality in chronic heart failure. Lancet. 1997 Apr 12;349(9058):1050-3. doi: 10.1016/S0140-6736(96)07015-8. PMID 9107242
- [Background] Mandic S, Myers J, Selig SE, Levinger I. Resistance versus aerobic exercise training in chronic heart failure. Curr Heart Fail Rep. 2012 Mar;9(1):57-64. doi: 10.1007/s11897-011-0078-0. PMID 22131070
- [Background] Zizola C, Schulze PC. Metabolic and structural impairment of skeletal muscle in heart failure. Heart Fail Rev. 2013 Sep;18(5):623-30. doi: 10.1007/s10741-012-9353-8. PMID 23065040
- [Background] Toth MJ, Miller MS, VanBuren P, Bedrin NG, LeWinter MM, Ades PA, Palmer BM. Resistance training alters skeletal muscle structure and function in human heart failure: effects at the tissue, cellular and molecular levels. J Physiol. 2012 Mar 1;590(5):1243-59. doi: 10.1113/jphysiol.2011.219659. Epub 2011 Dec 23. PMID 22199163
- [Background] Braith RW, Welsch MA, Feigenbaum MS, Kluess HA, Pepine CJ. Neuroendocrine activation in heart failure is modified by endurance exercise training. J Am Coll Cardiol. 1999 Oct;34(4):1170-5. doi: 10.1016/s0735-1097(99)00339-3. PMID 10520808
- [Background] Volaklis KA, Tokmakidis SP. Resistance exercise training in patients with heart failure. Sports Med. 2005;35(12):1085-103. doi: 10.2165/00007256-200535120-00006. PMID 16336010
- [Background] Cohen S, Nathan JA, Goldberg AL. Muscle wasting in disease: molecular mechanisms and promising therapies. Nat Rev Drug Discov. 2015 Jan;14(1):58-74. doi: 10.1038/nrd4467. PMID 25549588
- [Background] Meyer P, Gayda M, Juneau M, Nigam A. High-intensity aerobic interval exercise in chronic heart failure. Curr Heart Fail Rep. 2013 Jun;10(2):130-8. doi: 10.1007/s11897-013-0130-3. PMID 23397179
- [Background] Santa-Clara H, Fernhall B, Mendes M, Sardinha LB. Effect of a 1 year combined aerobic- and weight-training exercise programme on aerobic capacity and ventilatory threshold in patients suffering from coronary artery disease. Eur J Appl Physiol. 2002 Oct;87(6):568-75. doi: 10.1007/s00421-002-0675-4. Epub 2002 Jul 30. PMID 12355198
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Brown K. A review to examine the use of SF-36 in cardiac rehabilitation. Br J Nurs. 2003 Aug 14-Sep 10;12(15):904-9. doi: 10.12968/bjon.2003.12.15.11422. PMID 12937366
- [Background] Ferreira PL. [Development of the Portuguese version of MOS SF-36. Part I. Cultural and linguistic adaptation]. Acta Med Port. 2000 Jan-Apr;13(1-2):55-66. Portuguese. PMID 11059056

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT03320655/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT03320655/ICF_001.pdf